CLINICAL TRIAL: NCT03958864
Title: A PHASE 1, OPEN LABEL STUDY TO EVALUATE THE PHARMACOKINETICS AND SAFETY/TOLERABILITY OF CC-90001 IN JAPANESE HEALTHY SUBJECTS
Brief Title: A Study of Safety, Tolerability, and Pharmacokinetics of Multiple-Dose CC-90001 in Japanese and Caucasian Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-90001-CP-006; U1111-1229-5813
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteer
Keywords: Healthy Subjects; CC-90001; Japanese; Caucasian; Safety; Pharmacokinetics
MeSH Terms: interventions — CC-90001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CC-90001 100 mg (Experimental): 100 mg of CC-90001 (once daily [QD] x 7 days) will be given orally
  Interventions: Drug: CC-90001
- CC-90001 200 mg (Experimental): 200 mg of CC-90001 (once daily [QD] x 7 days) will be given orally
  Interventions: Drug: CC-90001
- CC-90001 400 mg (Experimental): 400 mg of CC-90001 (once daily [QD] x 7 days) will be given orally
  Interventions: Drug: CC-90001

INTERVENTIONS:
Drug: CC-90001 — CC-90001

SUMMARY:
This is a Phase 1, open-label, randomized, parallel design study to evaluate the PK and safety/tolerability of CC 90001 in Japanese and Caucasian healthy adult subjects.

The study will consist of multiple oral doses of IP (QD x 7 days) in 3 planned dose level cohorts of 100 mg, 200 mg, and 400 mg. Each cohort will have 20 subjects (10 Japanese subjects and 10 Caucasian subjects, with a minimum of 8 subjects to complete in each group) who will receive IP (see below).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be enrolled in the study:

1. Healthy, adult, male and female subjects.
2. Japanese subjects who were born in Japan and not have lived outside of Japan for more than 10 years, have both parents and grandparents of Japanese origin, and have not significantly modified their diets since leaving Japan.
3. Caucasian subjects who have age and body mass index matched with Japanese subjects.

Exclusion Criteria:

1. Has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study or place the subject at unacceptable risk if he/she were to participate in the study.
2. Use of any prescribed systemic or topical medication within 30 days of the first dose administration.
3. Has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, and excretion.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- AUC0-t | Day 1 and Day 7- 10
  Area under the plasma concentration-time curve from time zero to the time point of the last measurable concentration
Pharmacokinetic- AUC0-∞ | Day 1 and Day 7- 10
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetic- CL/F | Day 1 and Day 7- 10
  Estimation of apparent clearance of drug from plasma after extravascular administration
Pharmacokinetic- Vz/F | Day 1 and Day 7- 10
  Estimation of apparent volume of distribution during the terminal phase
Pharmacokinetic- Cmax | Day 1 and Day 7
  Estimation of observed maximum plasma concentration
Pharmacokinetic- Tmax | Day 1 and Day 7
  Estimation of time to Cmax
Pharmacokinetic- t1/2 | Day 1 and Day 7- 10
  Description: Estimation of terminal elimination half-life

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number participants with Adverse Event

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ye, PhD, Study Director — Celgene
Locations (1):
- Paraxel International, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/